CLINICAL TRIAL: NCT05898295
Title: Assessment of the Behavior of the Preterm Newborn: Discriminative and Predictive Capacity of the Sensory-motor Behavior Observation Grid
Brief Title: Assessment of the Behavior of the Preterm Newborns
Acronym: GOCSM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Cristina Borradori Tolsa, principal investigator, University Hospital, Geneva
Other Study IDs: ID 2020-00572
Record Dates: First submitted 2023-05-10; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Premature Birth
Keywords: premature birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — No intervention: only observation of the child behavior

SUMMARY:
The project presented here aims to evaluate the discrimination capacity of the Observation of Sensory-Motor Behavior (OSMB) grid of the preterm infant, as well as its predictive capacity for the child's later psychomotor development.

To do this, OSMB grids will be completed during dystimulant care and during stabilizing care in 65 preterm infants. In addition, an OSMB grid will also be completed during a sensorimotor assessment at 37 weeks gestational age and at 1 month corrected for prematurity in 100 preterm infants. The OCSM scores will then be compared to the Bayley III scale scores at 6 months of age corrected for prematurity.

DETAILED DESCRIPTION:
The project presented here aims to evaluate the discrimination capacity of the Observation of Sensory-Motor Behavior (OSMB) grid of the preterm infant, as well as its predictive capacity for the child's later psychomotor development.

To do this, OSMB grids will be completed during dystimulant care and during stabilizing care in 65 preterm infants. In addition, an OSMB grid will also be completed during a sensorimotor assessment at 37 weeks gestational age and at 1 month corrected for prematurity in 100 preterm infants. The OCSM scores will then be compared to the Bayley III scale scores at 6 months of age corrected for prematurity.

ELIGIBILITY:
Inclusion Criteria:

* <37weeks
* Hospitalized in Geneva Hospital NICU
* At least one parent speaking french

Exclusion Criteria:

* No exclusion cirteria

Ages: 3 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children born before 37+0/7 weeks of gestation and hospitalized in the NICU of Geneva hospitals are recruited. At least one French speaking parent is required to ensure parents understand the study.
  Children are recruited before 1 month of corrected age appointment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing the ability of the OSMB grid to discriminate the sensory-motor status of the preterm newborn in routine neonatal care practice | between birth and hospital discharge (up to 200days)
  Observation of the child's behavior during a disstimulating treatment and during a stabilizing treatment using the Observation of Sensory-Motor Behavior (OSMB) grid
To evaluate the predictive capacity of the child's later psychomotor development on the basis of the items from the sensorimotor assessment thanks to the OCSM grid, at term equivalent age | between 37 and 40weeks of gestational age
  Evaluation of newborns' development using the Observation of Sensory-Motor Behavior (OSMB) grid
To evaluate the predictive capacity of the child's later psychomotor development on the basis of the items from the sensorimotor assessment thanks to the OCSM grid, at term equivalent age | and 1 month of corrected age
  Evaluation of newborns' development using the Observation of Sensory-Motor Behavior (OSMB) grid

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Universitaire de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No